CLINICAL TRIAL: NCT05738915
Title: Role of C-Reactive Protein /Albumin Ratio in Evaluation of Disease Activity in Patients With Inflammatory Bowel Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Abd El Raheem, Role of C-Reactive Protein /Albumin Ratio in evaluation of Disease Activity in Patients with Inflammatory Bowel Disease, Assiut University
Other Study IDs: CRP/Albumin Ratio in IBD
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CRP/Albumin ratio in IBD — Role of C-Reactive Protein /Albumin Ratio in evaluation of Disease Activity in Patients with Inflammatory Bowel Disease.

SUMMARY:
Role of C-Reactive Protein /Albumin Ratio in evaluation of Disease Activity in Patients with Inflammatory Bowel Disease.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) is defined as a life long chronic inflammatory disease affecting the gastrointestinal tract resulting from the interaction of environmental and genetic elements, has been a global healthcare problem with a steadily increasing incide IBD is mainly composed of two different bowel-relapsing disorders, including Crohn's disease (CD) and ulcerative colitis (UC).

Early detection of the disease activity of IBD is of great significance for the treatment of this disease, which can effectively prevent complications and therefore improve prognosis as well as quality of life. In current clinical practice, commonly used noninvasive biomarkers such as C-reactive protein (CRP) and erythrocyte sedimentation rate (ESR), are considered to be important for both early diagnosis and accurate monitoring of the disease activity in IBD patients.

The C-reactive protein/albumin ratio (CAR) is indicative of the balance between inflammation and nutritional status, making it an excellent marker for assessing disease activity in patients The disease activity of UC and CD patients was evaluated by the Mayo score and Crohn disease activity inde (CDAI).

ELIGIBILITY:
Inclusion Criteria:

* patients with IBD which included Crohn disease and Ulcertive colitis patients above age 18 years old.

Exclusion Criteria:

* concurrent infections, liver cirrhosis, hematological diseases, heart failure, malignancies, autoimmune diseases, or congenital or acquired immunodeficiencies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - patients with IBD which included Crohn disease and Ulcertive colitis patients above age 18 years old.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02-15 (Estimated); Primary Completion 2023-07-15 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
CRP/Albumin ratio in IBD | Baseline
  Role of C-Reactive Protein /Albumin Ratio in evaluation of Disease Activity in Patients with Inflammatory Bowel Disease.